CLINICAL TRIAL: NCT01976221
Title: Priority Setting and Waiting Time Decision in the Referral Process, How and by Whom? A Prospective Cluster Randomized Controlled Trial on the Effects of an Education Program in Priority Setting and Waiting Time Decision in Referrals
Brief Title: Priority Setting and Waiting Time Decision in the Referral Process, How and by Whom?
Acronym: Priority
Status: Withdrawn | Type: Observational
Why Stopped: Study withdrawn
Sponsor: University of Bergen (Other)
Responsible Party: Principal Investigator, Olav Thorsen, MD, University of Bergen
Other Study IDs: REK2013/1762
Record Dates: First submitted 2013-10-17; First posted 2013-11-05 (Estimated); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Communication
Keywords: Comprehensive referrals; Appropriate referring; Priority setting; Waiting time in hospital
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prioritization: Team-based multifaceted interactive training

SUMMARY:
The referral letter is used for different purposes: a request for a special diagnostic assessment or medical treatment that the GP cannot perform for the patient, an invitation to have a second opinion about a clinical problem or a wish for mutual responsibility for the medical handling. The individual referral rate between GPs varies greatly, and is an important determinant of secondary care utilization. We wanted to study the various elements and factors having an impact on the referral process, from the moment the GP decides to refer the patient until the hospital consultant assess the referral and prioritise the patient for further investigation or treatment. How and why are we, the GPs who refer, so different? We wanted to

1. identify and describe general practitioners' reflections on and attitudes to the referral process and cooperation with hospital specialists
2. identify and describe hospital consultants' reflections on and attitudes to the referral process and cooperation with general practitioners
3. identify typologies characterising GPs in the referral practice

DETAILED DESCRIPTION:
Design and Methods:

We did two qualitative and one quantitative study. The first was a focus group study with GPs in CPD groups, the second an individual study with hospital consultants, both analyses by using systematic text condensation. The third was a quantitative registration of impressions, facts and feelings in the referral process using a principal component analysis to find typologies for GPs who refer to hospital.

Participants:

GPs referring to Stavanger University Hospital. Hospital consultants at Stavanger University Hospital.

Intervention: No intervention was performed.

Time schedule:

Data Collection finished May 2014.

ELIGIBILITY:
Inclusion Criteria:

All the 300 GPs referring to Stavanger University Hospital who participate in one of the 58 CPD groups in South Rogaland County and who agree to participate in the study are included.

Exclusion Criteria:

GPs not willing to participate

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General practitioners referring to Stavanger University Hospital
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2018-10-10 (Estimated)

PRIMARY OUTCOMES:
Use of priority setting and waiting time indication in referrals | 1 year
  The use of priority setting and waiting time in referrals will be recorded before and after an intervention with group training for general practitioners

SECONDARY OUTCOMES:
Referral rates | One year
  The referral rates may be reduced by higher awareness of non-prioritized medical conditions. The use of priority setting and waiting time according to the national prioritization guidelines can give a higher correlation between GPs and hospital consultants about priority setting and waiting time.

OTHER OUTCOMES:
Inter-rater agreement between GPs and hospital consultants on priority setting and waiting time for patients | One year
  We will study the inter-rater correlation between GPs and hospital consultants about priority setting and waiting time for patients referred to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anders Baerheim, Professor, Study Chair — Department of Global Public Health and Primary Care, University of Bergen, Norway
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thorsen O, Hartveit M, Baerheim A. General practitioners' reflections on referring: an asymmetric or non-dialogical process? Scand J Prim Health Care. 2012 Dec;30(4):241-6. doi: 10.3109/02813432.2012.711190. Epub 2012 Oct 10. PMID 23050793